CLINICAL TRIAL: NCT02148042
Title: Overgeneralization of Conditioned Fear as a Pathogenic Marker of Anorexia Nervosa
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1312M46141
Record Dates: First submitted 2014-05-20; First posted 2014-05-28 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Anorexia; Generalized Anxiety
Keywords: Anorexia; Generalized anxiety; Fear
MeSH Terms: conditions — Anorexia; Generalized Anxiety Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Anorexics
- Controls

SUMMARY:
Anorexia nervosa is a chronic mental health condition characterized by maladaptive food consumption (i.e., hypophagia) and distorted body image. There is substantial evidence of a phenotypic overlap between anorexia nervosa and anxiety disorders, as well as data suggesting the two share a common genetic pathway. Despite these findings, little research has examined fear conditioning among individuals with anorexia nervosa, and no research has examined whether individuals with anorexia nervosa have a propensity to overgeneralize conditioned fear stimuli, one of the more robust fear-conditioning markers of anxiety disorders. The current study assesses generalization of conditioned fear with fear-potentiated startle: the cross-species enhancement of the startle reflex when an organism is in a state of fear. Animal data, as well as an emerging literature in humans, tightly links fear-potentiated startle to the amygdala-based fear circuit. Thus, evidence of overgeneralized fear-potentiated startle in anorexia nervosa would link this eating disorder to hypersensitivity of the fear circuit and could inform the development of novel pharmacologic and psychological treatments for anorexia nervosa based on treatment models used in the anxiety disorders literature.

DETAILED DESCRIPTION:
The overarching objective of the current proposal is to examine the feasibility of applying a generalization of conditioned fear-potentiated startle paradigm, which has been used successfully to measure the sensitivity of fear networks in anxiety disorders, to adults with anorexia nervosa. The specific aim will be to examine whether conditioned-fear generalization gradients in anorexia nervosa participants differ from those in healthy controls. It is hypothesized that anorexia nervosa participants will display stronger generalization as indicated by less quadratic generalization gradients (i.e., a more gradual decline in conditioned fear as the generalization stimuli deviate from the conditioned fearful stimuli), which is indicative of a heightened sensitivity, or lower thresholds of activation, in the fear circuit (i.e., less danger information necessary to trigger the fear).

ELIGIBILITY:
Inclusion Criteria:

* Adults (age≥18)

  a. Anorexics
* Meet criteria for Diagnostic and Statistical Manual (DSM-5) anorexia nervosa

  b. Controls
* age matched
* sex-matched

Exclusion Criteria:

* Criteria are met for a current or past Axis I disorder.
* Inability to read English
* Pregnancy/lactation
* Acute suicidality
* Medical instability as determined by a medical history visit and serum electrolyte testing,
* Medical conditions that may place the participant at risk (e.g., cardiovascular condition)
* Current use of medication that alter central nervous system function

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Fifteen adults with anorexia nervosa and 15 healthy, age- and sex- matched control participants will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2014-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
The primary outcome variable is startle response (eye blink). | Within 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kelly C. Berg, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States